CLINICAL TRIAL: NCT02749019
Title: 68Ga-NOTA-BBN-RGD PET/CT in Breast Cancer Patients
Brief Title: Dual Integrin αvβ3 and GRPR Targeting PET Imaging in Breast Cancer Patients
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PUMCHNM012; ZIAEB000073 (NIH)
Record Dates: First submitted 2016-04-20; First posted 2016-04-22 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Breast Cancer
Keywords: BBN-RGD; GRPR; integrin αvβ3
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 68Ga-NOTA-BBN-RGD PET/CT (Experimental): The patients were injected with 111-148 MBq of 68Ga-NOTA-BBN-RGD in one dose intravenously and underwent PET/CT scan 15-30 min later.
  Interventions: Drug: 68Ga-NOTA-BBN-RGD

INTERVENTIONS:
Drug: 68Ga-NOTA-BBN-RGD — 68Ga-NOTA-BBN-RGD were injected into the patients before the PET/CT scans

SUMMARY:
This is an open-label positron emission tomography/computed tomography (PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-BBN-RGD in breast cancer patients. A single dose of 111-148 Mega-Becquerel (MBq) 68Ga-NOTA-BBN-RGD will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
Gastrin-releasing peptide receptor (GRPR) is a member of the G protein-coupled receptor family of bombesin receptors, which is over-expressed in various types of cancer cells, including prostate cancer, breast cancer, colorectal cancer, pancreatic cancer, glioma, lung cancer, ovarian cancers, endometrial cancers, renal cell cancer and gastrointestinal stromal tumors. BBN(7-14), with the amino acid sequence of Gln-Trp-Ala-Val-Gly-His-Leu-Met-NH2, has been extensively used for the development of molecular probes for the imaging of GRPR. On the other hand, the RGD moiety binds with integrin αvβ3 receptor, also plays an important role in the regulation of tumor growth, angiogenesis, local invasiveness, and metastatic potential in human breast cancer. To target both receptors, a heterodimeric peptide BBN-RGD was synthesized from bombesin(7-14) and c(RGDyK) through a glutamate linker and then labeled with 68Ga. An open-label whole-body PET/ CT study was designed to investigate the safety and dosimetry of 68Ga-NOTA-BBN-RGD and diagnostic performance of 68Ga-NOTA-BBN-RGD PET/CT in breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Neoplasm identified by X-ray, ultrasound or MRI as breast cancer
* To provide basic information and sign the written informed consent.

Exclusion Criteria:

* Consisted of conditions of mental illness;
* Severe liver or kidney disease with serum creatinine > 3.0 mg/dl (270 μΜ) or any hepatic enzyme level 5 times or more than normal upper limit;
* Severe allergy or hypersensitivity to IV radiographic contrast
* Claustrophobia to accept the PET/CT scanning
* Pregnancy or breast feeding

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-NOTA-BBN-RGD in breast cancer | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in breast cancer will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China